CLINICAL TRIAL: NCT06069401
Title: Microvascular Resistance Reserve Assessment Derived From Absolute Flow and Resistance by PET and CT
Brief Title: The MASTER-PACT Study
Acronym: MASTER-PACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Paul Knaapen, Prof. Dr. P. Knaapen, Amsterdam UMC, location VUmc
Other Study IDs: NL84769.018.23
Record Dates: First submitted 2023-09-20; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Microvascular Coronary Artery Disease; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to compare non-invasive myocardial perfusion reserve (MRR) to invasively measured MRR in patients suspected for coronary artery disease (CAD).

The main question it aims to answer is:

• what is the correlation and agreement between non-invasive and invasive MRR.

Participants suspected for CAD and referred for invasive coronary angiogram (ICA) will receive a [15O]H2O-PET and coronary CT angiography preceding ICA. During ICA, microvascular resistance measurements will be performed using thermodilution.

DETAILED DESCRIPTION:
Rationale:

In at least 25% - 50% of patients with chest pain, myocardial ischemia can be present without angiographic evidence of significant epicardial disease. In such patients, it is often assumed that the microvasculature of the myocardium is abnormal, called coronary microvascular dysfunction (CMD). This microvascular dysfunction constitutes a diagnostic and therapeutic problem with considerable morbidity and associated functional limitations, reduces quality of life, impairs outcome, and increases economic burden for healthcare systems. In the last years, a new invasive methodology has been developed for true quantitative investigation of the coronary microcirculation by calculation of the microvascular resistance reserve (MRR). Non-invasively, calculating the MRR is also possible by measuring resting and hyperemic myocardial blood flow (MBF), for example using quantitative Positron Emission Tomography (PET). However, non-invasive MRR can only be calculated by PET alone in the complete absence of any epicardial disease (i.e. a Fractional Flow Reserve [FFR] of 1.0). In order to obtain information on epicardial disease without using invasive interrogation of the coronary arteries, a method has been developed by HeartFlow Inc. to combine PET and FFR calculated from Coronary Computed Tomography Angiography (FFRCT). Using this method, MRR can be calculated non-invasively regardless of the presence of epicardial disease. However, non-invasive MRR has never been validated against invasively measured MRR.

Objective:

The main objective is to compare non-invasive MRR, obtained using PET and FFRCT (CT-scanning), with invasively measured MRR measurement using continuous thermodilution.

Study design:

This study is a prospective validation study in which all patients will undergo dual energy CCTA and [15O]H2O PET scan before invasive coronary angiography (ICA) in conjunction with invasive flow/pressure and thermodilution measurements.

Study population:

Chronic coronary syndrome patients without documented coronary artery disease (CAD) referred for ICA will be evaluated for inclusion.

Main study parameters/endpoints:

The primary endpoint will be the correlation and agreement between non-invasive and invasive MRR. To achieve our study objective, MRR calculated by PET and FFRCT will be compared to invasively measured MMR.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

A three day protocol will be completed after referral ensuring the diagnostic work-up of patients is not delayed. On day 1 patients will undergo CCTA. On day 2, patients will receive PET scan. Then, on day 3, irrespective of CCTA and PET results, patients will undergo ICA with invasive pressure/thermodilution measurements. The risks of CT and PET are considered to be low. Patients are referred for a clinically indicated ICA and as such risks of the ICA are not deemed study-related. The risk of invasive measurements during ICA are considered low. No direct benefit is present for the participating patients. Nevertheless, measurement of FFR, microvascular resistance and MRR is often useful to make a better decision on performing or deferring PCI, is helpful to better understand the nature of angina complaints in these patients, and contributes to fine-tuning of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Referred for ICA because of suspected CAD
2. No documented prior history of CAD
3. Age ≥18 and ≤80 years old

Exclusion Criteria:

1. Unstable CAD, Non-ST-Elevation Myocardial Infarction (NSTEMI), ST-Elevation Myocardial Infarction (STEMI), cardiogenic shock or hemodynamically unstable patients
2. Patients with previous coronary artery bypass (CABG) surgery, PCI or myocardial infarction (MI)
3. Tortuous or calcified coronary arteries, if known
4. Coronary arteries with a small caliber (<2,5 mm), if known
5. Atrial fibrillation, second or third degree atrioventricular block or severe conduction disturbances with an indication for temporary or permanent pacing
6. History of severe COPD or chronic asthma
7. Renal failure ( i.e. eGFR < 30 mL/min)
8. Use of sildenafil (Viagra) or dipyramidol (Persantin) that cannot be terminated
9. Contra-indications for β-blockers
10. Allergic reaction to iodized contrast
11. Pregnancy
12. Inability to understand and give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic coronary syndrome patients without documented coronary artery disease (CAD) referred for ICA will be evaluated for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation non-invasive and invasive MRR | Immediately after the PET and CT scan (non-invasive MRR) and ICA (invasive MRR)
  The first primary endpoint will be correlation between non-invasive and invasive MRR, indicated by Pearson/Spearman correlation.
Agreement non-invasive and invasive MRR | Immediately after the PET and CT scan (non-invasive MRR) and ICA (invasive MRR)
  The first primary endpoint will be agreement between non-invasive and invasive MRR, indicated by a Blant-Altman analysis.

SECONDARY OUTCOMES:
Correlation non-invasive and invasive resting and hyperemic resistance | Immediately after the PET and CT scan (non-invasive MRR) and ICA (invasive MRR)
  The first secondary endpoint will be correlation between non-invasively and invasively measured resting and hyperemic resistance, indicated by Pearson/Spearman correlation.
Agreement non-invasive and invasive resting and hyperemic resistance | Immediately after the PET and CT scan (non-invasive MRR) and ICA (invasive MRR)
  The first secondary endpoint will be agreement between non-invasively and invasively measured resting and hyperemic resistance, indicated by a Blant-Altman analysis.

IPD SHARING:
Plan to Share IPD: No